CLINICAL TRIAL: NCT07365696
Title: Fatigue Och Kognitiv Dysfunktion Till följd av Synaptopati Eller Graft Versus Host (GVH) Sjukdom i hjärnan.
Brief Title: Fatigue and Cognitive Dysfunction Due to Synaptopathy or Graft Versus Host (GVH) Disease in the Brain.
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ksenia Boriskina, MD, Karolinska University Hospital
Other Study IDs: 2023-02021-01
Record Dates: First submitted 2023-11-27; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Graft Vs Host Disease; Cognitive Dysfunction
MeSH Terms: conditions — Fatigue; Graft vs Host Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with fatigue and cognitive dysfunction
  Interventions: Radiation: PET investigation
- Patients without fatigue and cognitive dysfunction
  Interventions: Radiation: PET investigation

INTERVENTIONS:
Radiation: PET investigation — Trial subjects will undergo two advanced PET investigations

SUMMARY:
Patients undergoing allogenic stem cell transplantation are regularly followed up in the outpatient clinic at Karolinska University Hospital. Here, patients are offered participation the fatigue study measuring both fatigue and cognitive impairment systematically by international standard. Meanwhile liquor samples and advanced PET imaging techniques are available for these patients as part of a research project allowing extensive immunological and radio-morphological studies.

ELIGIBILITY:
Inclusion Criteria: PET images available retrospectively

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergone allogeneic stemcell transplantation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
To investigate the role of inflammation on synaptic density and glial cell activation as the cause of mental fatigue and cognitive dysfunction in survivors after alloSCT. | 2024-2027
  Analysis of PET imaging (both descriptive and radiokinetical) in combination with biological markers for neuroinflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ksenia Boriskina, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No